CLINICAL TRIAL: NCT03369626
Title: Effectiveness of a Digital Therapeutic in a Geographically Distributed Population With Type 2 Diabetes
Brief Title: Effectiveness of a Digital Therapeutic on Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FareWell (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: dmstudyv4
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Intervention Model Description: evaluation of pre/post measures of a single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FareWell Program (Other): All participants receive the FareWell Program intervention in this evaluation study
  Interventions: Behavioral: FareWell Program

INTERVENTIONS:
Behavioral: FareWell Program — The FareWell Program is a digitally delivered lifestyle management curriculum, which includes meal planning tools, daily self monitoring, personalized goal setting and bi-weekly live one-on-one health coaching.

SUMMARY:
A clinical study evaluating a three month digitally delivered lifestyle change program in adults with Type 2 Diabetes. The FareWell Program (the "Program") aims to reduce well-established biomarkers of cardiometabolic diseases, weight, and medications. The current study is designed to evaluate to what degree adults with Type 2 Diabetes engaged with the Program can improve glycemic control and/or decrease medication needs.

DETAILED DESCRIPTION:
The Program aims to reduce well-established biomarkers of cardiometabolic diseases, weight, and medications. It includes meal planning tools, smart shopping lists, recipes curated by a physician, dietitian and chef educator, daily self-monitoring features with personalized weekly goals, bi-weekly live one-on-one health coaching and support from an online member community, and an educational curriculum. Subjects in the Program may receive support from other members of a Care Team (lifestyle medicine physician, chef educator, registered dietitian and/or psychologist/psychiatrist) as needed. The Care Team does not provide medical advice, nor replace traditional medical care. Instead, the Care Team encourages behavior change by providing support and sharing its expertise.

Study participants will have access to the Program for a twelve week period and will be asked to complete short health surveys at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes

Exclusion Criteria:

* Inability to understand, consent to, or comply with the study protocol for any reason, including inability to read or comprehend English.
* Does not have a smartphone (either an iPhone or Android phone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Level of engagement with the assigned mobile app | 12 weeks
  How do participants interact with the digital program (e.g. feature use, coaching calls completed, targets tracked, targets met)

SECONDARY OUTCOMES:
Change in self-reported Hemoglobin A1c | 12 weeks
  Comparison of baseline and end program self reported Hemoglobin A1c
Change in self-reported diabetes medication type or dose | 12 weeks
  Comparison of diabetes medications reported at baseline to any changes reported at the end of the study or mid-study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Berman, MD, Principal Investigator — FareWell
Locations (1):
- FareWell LLC, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided